CLINICAL TRIAL: NCT06956417
Title: REhabilitation of MEMory Symptoms After BRain Concussion
Acronym: REMEMBR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H24-02486
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Concussion, Brain; Mild Traumatic Brain Injury
Keywords: Functional cognitive disorder
MeSH Terms: conditions — Brain Concussion | interventions — Cognitive Behavioral Therapy; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy
- Cognitive rehabilitation (Active Comparator)
  Interventions: Behavioral: Cognitive rehabilitation
- Waitlist - Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy (CBT) is delivered by a psychologist over 10 individual (1:1) manualized videoconference sessions. The goal of this therapy is for participants to use their memory more normally (i.e., reduce avoidance and safety behaviors) and view memory lapses as less threatening.
  Arms: Cognitive behavioral therapy
Behavioral: Cognitive rehabilitation — Cognitive compensatory strategy training (CCST), a traditional cognitive rehabilitation intervention, is delivered by a Occupational Therapist over 10 individual (1:1) manualized videoconference sessions. Participants optimize their use of current compensatory strategies and/or learn new ones suited to their needs and lifestyle. The goal is to minimize memory lapses in daily life.
  Arms: Cognitive rehabilitation

SUMMARY:
Persistent memory symptoms after concussion are common, and likely perpetuated by unhelpful illness beliefs and coping behaviors. Results from a pilot study suggested that traditional cognitive rehabilitation and a novel cognitive-behavioral therapy (CBT) protocol were both associated with improvements in subjective memory functioning. The present study will more definitively compare the effectiveness of these interventions for improving subjective memory functioning after concussion.

DETAILED DESCRIPTION:
The primary research aims of this study are to determine whether cognitive behavioral therapy (CBT) and cognitive compensatory strategy training (CCST) improves subjective memory functioning compared to usual care, and to compare the effectiveness of CBT and CCST. This study is a multisite three-armed randomized control trial (RCT) that will randomize adults with persistent memory symptoms following concussion to CBT, CCST, or a covert waitlist condition (2:2:1). Participants will be blinded to the other arms of the study and the study hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-59
2. Concussion diagnosis confirmed with structured interview based on American Congress of Rehabilitation Medicine diagnostic criteria
3. Concussion occurred between 6 and 36 months before enrollment
4. Ongoing memory concerns
5. Fluent in English
6. Stable access to a computer, tablet, or smartphone with internet capability

Exclusion Criteria:

1. Fail performance validity testing
2. Comorbid psychiatric or neurological disorder or is taking a medication that could fully account for their memory symptoms

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Multifactorial Memory Questionnaire-Satisfaction scale | Week 20
  Measures participants' concern, satisfaction, and overall appraisal of their memory ability. Participants rate their agreement with 18 statements. Total scores range from 0 to 72, with lower total scores indicating worse subjective memory functioning.

SECONDARY OUTCOMES:
Fear-Avoidance of Memory Loss Scale | Week 1 and week 20
  Assesses fears and avoidance behaviors associated with memory decline. Participants rate 24 items on a 5-point scale, where the higher scores indicate greater memory concern and maladaptive coping.
Patient Global Impression of Change scale | Week 20
  Participants rate how much their memory functioning has improved or declined overall since the beginning of the study, on a single item rated on a 7-point scale where the midpoint is no change.
Work and Social Adjustment Scale | Week 1 and week 20
  Participants rate how much their condition interferes with their ability to carry out occupational and social activities across 5 items, on a scale from 1-7 where higher scores indicate more difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Noah D Silverberg, PhD, Principal Investigator — University of British Columbia
Locations (9):
- Canada (9):
  - Calgary Brain Injury Program, Calgary, Alberta
  - Fraser Health Acquired Brain Injury and Concussion Services, Langley, British Columbia
  - G.F. Strong Adult Concussion Services, Vancouver, British Columbia
  - Integrated Adult Concussion Program at Hamilton Health Sciences, Hamilton, Ontario
  - 360 Concussion Care Clinic, Ottawa, Ontario
  - Sunnybrook Traumatic Brain Injury Clinic, Toronto, Ontario
  - Head Injury Clinic at St. Michael's Hospital, Toronto, Ontario
  - Hull-Ellis Concussion and Research Clinic at University Health Network, Toronto, Ontario
  - Canadian Concussion Centre at Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rioux M, Mamman R, Byworth MT, Panenka WJ, Howard AK, Perez DL, Schmidt J, Courchesne C, LeMoult J, Heran MK, Silverberg ND. Pilot feasibility randomised controlled trial of cognitive-behavioural therapy for functional cognitive disorder after concussion. BMJ Neurol Open. 2024 Oct 11;6(2):e000666. doi: 10.1136/bmjno-2024-000666. eCollection 2024. PMID 39410977